CLINICAL TRIAL: NCT04234594
Title: A Randomized, Double-blind and Single-dose Study to Compare the Pharmacokinetic and Safety of QL1203 and Vectibix® in Healthy Male Subjects.
Brief Title: Comparing the Pharmacokinetic and Safety of QL1203 and Vectibix® in Healthy Males.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QL1203-002
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-01

CONDITIONS: Healthy Males
MeSH Terms: interventions — Panitumumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL1203 (Experimental): Participants only receive QL1203, 6mg/kg on Day 1.
  Interventions: Drug: QL1203
- Vectibix® (Active Comparator): Participants only received Vectibix®，6 mg/kg on Day 1.
  Interventions: Drug: Vectibix®

INTERVENTIONS:
Drug: QL1203 — 6 mg/kg intravenous (IV) infusion only once，on the first day.
  Arms: QL1203
Drug: Vectibix® — 6 mg/kg intravenous (IV) infusion only once，on the first day.
  Arms: Vectibix®

SUMMARY:
A randomized, double-blind and parallel group study to compare the pharmacokinetic and safety of QL1203 and Vectibix® in healthy males.

DETAILED DESCRIPTION:
This is a phase I,single center, randomized, double-blind，single-dose and parallel group clinical trial . The primary objective is to assess the pharmacokinetic similarity of of QL1203 or Vectibix® in healthy male volunteers. The secondary objective are to assess the Clinical safety and immunogenicity similarity of QL1203 or Vectibix® in healthy male volunteers".

ELIGIBILITY:
Inclusion Criteria:

* Subjects sign the informed consent form and fully understand purpose, nature, process and possible adverse reactions of the study, and are able to complete the study according to the study plan requirements.
* Male,18 years to 65 years of age.
* Weight ≧50.0 kg; body mass index (BMI) in the range of 19.0～ 26.0 kg / m^2.
* Subjects have no history of chronic diseases or serious diseases such as cardiovascular, liver, kidney, respiratory, blood and lymph, endocrine, immune, psychiatric, nervous, gastrointestinal system diseases and the general health is good.
* Clinical laboratory examination, chest X-ray, abdominal B-ultrasound, electrocardiogram, physical examination, vital signs and various examinations are normal or abnormal without clinical significance.

Exclusion Criteria:

* Subjects have used any biological product within 3 months prior to receiving the study drug, or have used any monoclonal antibody drugs within 9 months.
* Subjects have anallergic history to study drug or any drug component; or persons with allergic history to two or more drugs and food.
* Subjects have a history of interstitial lung disease.
* Subjects have a history of keratitis or long-term wearing of contact lens.
* Subjects have used any prescription drugs, over-the-counter medicines, Chinese herbal medicines, and vitamins within 2 weeks before receiving the study drugs.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC0-t ) | 36 days
  Area under the plasma concentration-time curve (AUC0-t ) from 0 o'clock to the last measurable concentration acquisition time t.

CONTACTS AND LOCATIONS:
Overall Officials: Weiwei Ouyang, Professor, Principal Investigator — Cancer Hospital of Guizhou Province
Locations (2):
- China (2):
  - Guizhou Cancer Hospital, Guiyang, Guizhou
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan